CLINICAL TRIAL: NCT03646201
Title: Reducing Solid Fat and Added Sugar Intakes in Low-income Preschoolers Through Environmental and Behavioral Portion Size Strategies
Brief Title: Feeding, Fun, and Families Study
Acronym: FFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USDA-310138; USDA AFRI 2011-68001-30148 (Other Grant/Funding Number: USDA National Institute of Food and Agriculture, AFRI)
Record Dates: First submitted 2017-01-17; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Childhood Obesity
Keywords: childhood; obesity; nutrition; intervention; portion size; behavioral; environmental; feeding practices
MeSH Terms: conditions — Pediatric Obesity; Obesity; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FFF (Experimental): FFF teaches authoritative parenting skills for reducing children's exposure to and intakes of SoFAS, including changes to the family food environment, mothers' own eating behaviors, and food parenting practices.
  Interventions: Behavioral: FFF
- Control Group (No Intervention): Data are collected at baseline and post intervention session.

INTERVENTIONS:
Behavioral: FFF — FFF teaches authoritative parenting skills for reducing children's exposure to and intakes of SoFAS, including changes to the family eating environment, mothers' own eating behaviors, and food parenting practices.
  Arms: FFF

SUMMARY:
To develop and evaluate the efficacy of Feeding Fun and Families (FFF), a nutrition education intervention for low-income mothers emphasizing authoritative food parenting skills, on preschool aged children's energy intakes from solid fats and added sugars (SoFAS), using a randomized controlled trial conducted in a clinic-based setting.

FFF will result in lower child SoFAS intakes compared to a no-treatment control group at the end of the 12 week intervention (primary outcome), adjusted for baseline values.

DETAILED DESCRIPTION:
Feeding Fun and Families (FFF) taught mothers authoritative parenting skills for reducing children's exposure to and intake of daily energy from SoFAS. FFF was developed and rigorously testing a contextually sensitive, state-of-the art nutrition education program for low-income mothers emphasizing parenting skills. This project represents the first systematic research to translate, from bench-to-bedside, the basic behavioral science on child portion size to clinic-based and then community level nutrition education programming. FFF is a nutrition education intervention emphasizing the "hows" of parenting around feeding young children. Authoritative parenting strategies will target the family food environment, mothers' own eating behaviors, and their child feeding practices. Based on previous research, strategies will attempt to reduce SoFAS portions offered to children by reducing the size of dishware (e.g. cups, bowls, plates) used to serve children and used by children to eat, reducing portion sizes of amorphous (e.g. pasta) and unit foods (e.g. juice box) served to children, and encourage feeding practices that provide structure and autonomy support. The primary outcome, measured at baseline and at the end of the 12 week intervention, children's energy intake of discretionary calories from SoFAS.

Formative qualitative research was used to guide the development of FFF in a manner consistent with low-income mothers' parenting goals and responsive to their socioeconomic constraints. The FFF intervention was tested the "proof of concept" (i.e. efficacy) by evaluating an intensive version of the intervention in a randomized clinical trial (RCT). The findings were used to translate FFF for delivery by Supplemental Nutrition Assistance Program Education (SNAP-Ed) educators in urban communities of VA (VA), with the potential of being disseminated nationwide through the SNAP-Ed program.

Specific objectives were:

1. Phase I: Qualitatively understand the contextual factors (i.e. psychosocial, economic, structural) that will support mothers' acceptance and implementation of environmental and behavioral portion size strategies to decrease SFAS portions among low-income, at-risk preschoolers.
2. Phase II: To develop and evaluate the efficacy of the FFF obesity prevention nutrition education program for low-income mothers of preschoolers emphasizing behavioral and environmental parenting strategies around portion size in a clinic-based setting.

   • FFF will result in lower child SoFAS intakes compared to a no-treatment control group at the end of the 12 week intervention (primary outcome), adjusted for baseline values
3. Phase III: To translate the FFF program for delivery in SNAP-ED to mothers of preschool aged children.

ELIGIBILITY:
Inclusion Criteria:

* has a child that is 3-5 y at enrollment (up to 66 mo)
* Supplemental Nutrition Assistance Program (SNAP) eligible
* 18 y or older
* self-reported comfort with spoken and written English

Exclusion Criteria:

* child has a restrictive diet
* child has a severe food allergies
* child has a chronic illness or medication that influences intake/growth
* sever psychosocial impairment
* non-English speakers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-07; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Children's combined energy intake from solid fat and added sugars | At end of the FFF intervention (12 weeks), controlling for baseline values
  Daily intake (kcal/d); mean of 3, 24-hour dietary recalls. Recalls were administered using Nutrition Data System for Research Software by trained and certified staff at the Nutrition Coordinating Center (NCC), University of Minnesota, Minneapolis, MN who were blind to condition assignment.

SECONDARY OUTCOMES:
Children's total daily energy intake | At end of the FFF intervention (12 weeks), controlling for baseline values
  Daily intake (kcal/d); mean of 3, 24-hour dietary recalls. Recalls were administered using Nutrition Data System for Research Software by trained and certified staff at the Nutrition Coordinating Center (NCC), University of Minnesota, Minneapolis, MN who were blind to condition assignment.
Children's total daily solid fat intake | At end of the FFF intervention (12 weeks), controlling for baseline values
  Daily intake (kcal/d); mean of 3, 24-hour dietary recalls. Recalls were administered using Nutrition Data System for Research Software by trained and certified staff at the Nutrition Coordinating Center (NCC), University of Minnesota, Minneapolis, MN who were blind to condition assignment.
Children's total daily added sugar intake | At end of the FFF intervention (12 weeks), controlling for baseline values
  Daily intake (kcal/d); mean of 3, 24-hour dietary recalls. Recalls were administered using Nutrition Data System for Research Software by trained and certified staff at the Nutrition Coordinating Center (NCC), University of Minnesota, Minneapolis, MN who were blind to condition assignment.
BMI status | At end of the FFF intervention (12 weeks), controlling for baseline values
  Child height (cm) and weight (kg) will be measured in triplicate and converted to Body Mass Index z-scores specific to age and sex using Centers for Disease Control reference data.
Meal Observation | At the end of the FFF intervention (12 weeks)
  Nine maternal FFF target behaviors were observed at a buffet-style meal where mothers ate with their children. Mothers were assigned a total score representing the sum of target behaviors observed (possible score 0-9)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer O Fisher, Ph.D, Principal Investigator — Temple University
Locations (1):
- Temple University- Center for Obesity Research and Education, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herman AN, Malhotra K, Wright G, Fisher JO, Whitaker RC. A qualitative study of the aspirations and challenges of low-income mothers in feeding their preschool-aged children. Int J Behav Nutr Phys Act. 2012 Nov 16;9:132. doi: 10.1186/1479-5868-9-132. PMID 23157723
- [Background] Malhotra K, Herman AN, Wright G, Bruton Y, Fisher JO, Whitaker RC. Perceived benefits and challenges for low-income mothers of having family meals with preschool-aged children: childhood memories matter. J Acad Nutr Diet. 2013 Nov;113(11):1484-1493. doi: 10.1016/j.jand.2013.07.028. PMID 24144074
- [Background] Fisher JO, Wright G, Herman AN, Malhotra K, Serrano EL, Foster GD, Whitaker RC. "Snacks are not food". Low-income, urban mothers' perceptions of feeding snacks to their preschool-aged children. Appetite. 2015 Jan;84:61-7. doi: 10.1016/j.appet.2014.09.007. Epub 2014 Sep 18. PMID 25240637
- [Derived] Fisher JO, Serrano EL, Foster GD, Hart CN, Davey A, Bruton YP, Kilby L, Harnack L, Ruth KJ, Kachurak A, Lawman HG, Martin A, Polonsky HM. Title: efficacy of a food parenting intervention for mothers with low income to reduce preschooler's solid fat and added sugar intakes: a randomized controlled trial. Int J Behav Nutr Phys Act. 2019 Jan 17;16(1):6. doi: 10.1186/s12966-018-0764-3. PMID 30654818